CLINICAL TRIAL: NCT04119921
Title: Short-term Additive Effect of Topical Ketorolac on the Management of Diabetic Macular Edema With Intravitreal Bevacizumab
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 97377
Record Dates: First submitted 2019-10-02; First posted 2019-10-09 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2019-10

CONDITIONS: DME

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- usage of topical ketorolac in group1 (Active Comparator): usage of topical ketorolac every 6 hour in the first interval and then artificial tear every 6 hour as a placebo in the second interval.
  Interventions: Drug: prescription topical ketorolac in group 1
- usage of artificial tear in group 2 (Active Comparator): usage of artificial tear every 6 hour in the first interval and then topical ketorolac every 6 hour as a placebo in the second interval.
  Interventions: Drug: prescription artificial tear in group 2
- usage of artificial tear in group 1 (Active Comparator): usage of topical ketorolac every 6 hour in the first interval and then artificial tear every 6 hour as a placebo in the second interval
  Interventions: Drug: prescription artificial tear in group1
- usage of topical ketorolac in group2 (Active Comparator): usage of artificial tear every 6 hour in the first interval and then topical ketorolac every 6 hour as a placebo in the second interval
  Interventions: Drug: prescription topical ketorolac in group 2

INTERVENTIONS:
Drug: prescription topical ketorolac in group 1 — topical ketorolac every 6 hour in the first interval and then artificial tear every 6 hour as a placebo in the second interval.
  Arms: usage of topical ketorolac in group1
Drug: prescription artificial tear in group 2 — artificial tear every 6 hour in the first interval and then topical ketorolac every 6 hour as a placebo in the second interval.
  Arms: usage of artificial tear in group 2
Drug: prescription topical ketorolac in group 2 — artificial tear every 6 hour in the first interval and then topical ketorolac every 6 hour as a placebo in the second interval.
  Arms: usage of topical ketorolac in group2
Drug: prescription artificial tear in group1 — topical ketorolac every 6 hour in the first interval and then artificial tear every 6 hour as a placebo in the second interval.
  Arms: usage of artificial tear in group 1

SUMMARY:
Purpose: To evaluate the short-term effect of adding topical ketorolac to the management of diabetic macular edema (DME) with intravitreal bevacizumab (IVB).

Setting: Ophthalmology department of Imam Hossein and Torfe Medical Centers. Ophthalmic Epidemiology Research Center of Shahid Beheshti University of Medical Sciences Methods: In a randomized double-masked placebo-controlled crossover clinical trial, all eyes with DME with best-corrected visual acuity (BCVA) between 20/40 and 20/400 were included. They should have had at least one intravitreal anti-VEGF injection in the past 2 months. They were randomized into two groups. Both groups received two IVB injections with 6-week interval. One group received topical ketorolac every 6 hour in the first interval and then artificial tear every 6 hour as a placebo in the second interval. The other group received the opposite medications. Best-corrected visual acuity (BCVA) and central macular thickness (CMT) evaluations were repeated at the termination of each treatment period i.e. at 6 and 12 weeks. The main outcome measure was BCVA changes in logMAR and the second outcome was CMT changes. The interim analysis of this study is presented in this report.

ELIGIBILITY:
Inclusion Criteria:

* BCVA≤20/40 and BCVA 20/400 and better
* History of at least 1 intra-viteral bevacizumab (IVB) in the last 2 months
* Requires 2 IVB in the next 12 weeks
* Macular thickness >300 μm
* NO Other eye diseases
* Media clarity , pupillary dilation, and subject cooperation sufficient for adequate fundus photographs

Exclusion Criteria:

* hgb A1c> 8
* high risk PDR
* Macular edema due to a cause other than diabetic retinopathy
* Any other ocular condition that visual acuity would not improve from resolution of edema (eg.foveal atrophy)
* Prior treatment with intravitreal or peribulbar corticosteroid injection during last 3months
* History of macular photocoagulation during the last 6 months
* intraocular surgery(except cataract surgery)
* Cataract extractionin less than 6 months ago
* Uveitis ,NVG ,exudative AMD, HR PDR.
* Uncontrolled glaucoma
* Vitreomacular traction or epiretinal membrane

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
visual acuity | 6 weeks
  Snellen E-chart

SECONDARY OUTCOMES:
Centeral macular thickness | 6 weeks
  Ophtical Cohearence Tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran